CLINICAL TRIAL: NCT05065723
Title: Investigation of the Effect of Internet Addiction Level on Thumb Pressure Pain Threshold, Hand Strength and Manual Dexterity in University Students
Brief Title: Investigation of the Effect of Internet Addiction Level in University Students
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant Professor, Bandırma Onyedi Eylül University
Other Study IDs: AkcayB
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: University Students
Keywords: Internet Addiction; Pain Threshold; Hand Strength; Manual Dexterity
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The internet, which has become a part of our daily life; serves many purposes such as quick access to information, e-mail, and chat, banking and shopping, having a good time, using social networking sites. Internet addiction, which was first defined by Ivan Goldberg in 1996, is defined as the inability to control internet use, which causes pressure, feelings of anxiety, and dysfunctional behaviors in daily life activities. Social media, digital games and smartphone addiction are among the addiction types whose active ingredient is the internet, and internet addiction is expressed as a whole, regardless of the type of addictive application or activity. Considering that internet use is common among young people, one of the risk groups in terms of internet addiction is university students. As a matter of fact, Günay et al. stated that approximately 8% of university students are at risk of internet addiction.

In the literature, musculoskeletal problems and pain in the thumb and related joints, reduction in pinch strength, and hand function have been reported with smartphone use. In addition, a significant relationship was found between the time spent surfing the Internet and pain at the base of the thumb. However, to the best of our knowledge, no study has been found that examines the effect of internet addiction level on thumb pain threshold, hand strength and manual dexterity in university students. The aim of our research is to determine the level of internet addiction in university students and to examine the effect of internet addiction level on thumb pressure pain threshold, hand strength and manual dexterity.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being a student at Bandırma Onyedi Eylül University
* Willingness to participate in the study

Exclusion Criteria:

* Any injury involving the upper extremity in the last 6 months
* Any surgical operation involving the upper extremity in the last 6 months
* Any systemic disease
* Any neurological problems
* Use of any psychiatric medication

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students aged between 18-25 and studying at Bandırma Onyedi Eylül University
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Test | Baseline
  It was developed by Young and its Turkish validity and reliability study was performed by Bayraktar in 2001. The test consists of 20 items in total and is evaluated with a 6-point Likert type scale. In the test, which is scored between 0-100, people who score 49 or less are grouped as "No Symptom", people who score between 50 and 79 "Limited Symptom" and people who get 80 points or more are grouped as "Pathological Internet Users"
Pressure Pain Threshold | Baseline
  Pressure pain threshold, defined as the minimum force that triggers pain, is measured with an instrument called an algometer. The value obtained when the person indicates when the pressure sensation turns into a painful sensation is recorded in kg/cm²
Hand Strength | Baseline
  For the standard grip strength measurement, the person is asked to squeeze the dynamometer strongly and leave it completely loose while the elbow is in 90⁰ flexion and the forearm is in the neutral position, which is the standard test position of the American Hand Therapists Association, with a hand dynamometer. The average of the values obtained by measuring in 3 repetitions on the right and left hands is taken
Pinch Strength | Baseline
  The average is taken by measuring the pinchmeter in 3 repetitions on the right and left hands. In measurements, pinching force is evaluated by measuring in pinch, lateral and tripod grip positions
Minnesota Manual Dexterity Test | Baseline
  Black and red discs are used for Minnesota Manual Dexterity Test and it consists of 2 sub-parameters as Placement Test and Turning Test. The test measures gross dexterity, coordination, and speed
Purdue Pegboard Test | Baseline
  Developed by Tiffin in 1948; Its use in industrial candidates, veterans, college students, and people seeking vocational guidance has yielded important information about its validity and reliability, and practical implications. For the Purdue Peg Board Test, a platform consisting of two 0.45x0.29 m vertical columns, 25 test boards with 3 mm diameter holes in each, and 4 compartments containing pins (pegs), washers and collars is used. The test that evaluates fine dexterity unilaterally and bilaterally; It consists of a total of 4 subtest sections: Right Placement, Left Placement, Bilateral Placement and Right+Left+Bilateral Placement

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No